CLINICAL TRIAL: NCT02019511
Title: Safety Aspects of High-Dose Methylprednisolone in Fast-track Total Knee Arthroplasty
Brief Title: Safety Study of High-dose Methylprednisolone in Fast-track Total Knee Arthroplasty
Status: Withdrawn | Type: Observational
Why Stopped: The study design was too complex regarding aquisition of registry data.
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Lundbeck Foundation Centre for Fast-track Hip and Knee Arthroplasty (Unknown)
Responsible Party: Principal Investigator, Christoffer Joergensen, MD, Rigshospitalet, Denmark
Other Study IDs: RH-0703
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Infection of Total Knee Joint Prosthesis
Keywords: Orthopedic surgery; Infections; Steroid; Fast-track; Total knee arthroplasty; Safety
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- High dose Steroid: Patients scheduled for primary unilateral elective TKA Age >17 years
  none of the following contraindications for Methylprednisolone:
  * Allergy against Methylprednisolone.
  * Currently in systemic treatment with glucocorticoid
  * Current gastric ulcer
  * Insulin dependent diabetes mellitus
  Citizens without Danish social security number are not eligible for this study as follow-up is not possible.
- Historical cohort: Patients having primary unilateral elective TKA before initiation of Methylprednisolone as standard treatment
  age >17 years, Danish social security number
  and none of the following at time of surgery:
  * systemic treatment with glucocorticoid defined as: regular prescriptions on glucocorticoid within 2 months prior to surgery.
  * gastric ulcer defined as: prescriptions on drugs used in "triple therapy" for Helicobacter Pylori infection or prescriptions on antiacids/proton pump inhibitors beginning 1 month before surgery
  * Insulin dependent diabetes mellitus defined as: any prescriptions on insulin within 6 months prior to surgery
- Procedures without Steroid: Patients scheduled for primary unilateral elective TKA and age >17 years but who did not receive high dose Methylprednisolone regardless of reason.

SUMMARY:
It has been shown that a single high dose of steroid before surgery may reduce pain the first 48 hours after insertion of a new joint in the knee, a so called "total knee arthroplasty" (TKA). Consequently, this has been introduced as standard treatment of most patients at several Danish orthopedic departments. Although there are some concerns about the possibility of increased risk of prosthesis infections, this has not been proved in previous studies. However the studies are few, have limited number of patients and are not done using a standardized perioperative set-up.

This study is made to monitor the safety of a single high dose steroid injection before TKA, with regards to prosthesis infection within one year of surgery.

We hypothesize that there will be no increase in infections in patients receiving steroid injection before TKA compared to a historical cohort of patents who did not receive a steroid injection before their TKA.

DETAILED DESCRIPTION:
In order to reduce pain intensity as much as possible after surgical procedures, modern multimodal analgesic strategies using different analgetics targeting different mechanism of the pain reception system are used. At the same time this may reduce the use of opioids, which commonly cause sideeffects such as nausea, vomiting, obstipation,urinary retention, itching, respiratory suppression and sedation.

In spite of the use of a wide perioperative multimodal analgesia, pain after total knee arthroplasty (TKA), is stil a considerable clinical problem and need for optimisation of the immediate postoperative pain treatment. There is evidence that "high"dose glucocorticoids administered preoperatively reduces the level of pain and the use of opioids after surgery. A recent review did not give cause for concern regarding use of glucocorticoids in TKA,but found that data on longterm safety aspects are lacking, why no recommendations could be made.

As the limited evidence presently points to af benefit of glucocorticoids without serious side effects, the treatment has been introduced as standard treatment in TKA at several of the departments participating in the Lundbeck Foundation Centre for fast-track Hip and Knee Replacement collaboration.

This study is made to monitor the safety of high dose steroid injection before TKA, with regards to prosthesis infection within one year of surgery.

We hypothesize that there will be no increase in infections in patients receiving steroid injection before TKA compared to a historical cohort of patents who did not receive a steroid injection before their TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary unilateral elective TKA and no contraindications for high-dose Methylprednisolone preoperatively
* Danish Social security number

Exclusion Criteria:

One of the following contraindications for Methylprednisolone:

* Allergy against Methylprednisolone.
* Currently in systemic treatment with glucocorticoid
* Current gastric ulcer
* Insulin dependent diabetes mellitus

Further contraindications are at the discretion of the individual department/surgeon. The cohort without preoperative Methylprednisolone treatment will be followed as a separate cohort to identify potential selection bias.

- Citizens without Danish social security number are not eligible for this study as follow-up is not possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive unselcted patients with unilateral elective total fast-track knee arthroplasty in a standardized perioperative set-up and with completed prospective registration of preoperative chartacteristics and co-morbidity
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
prosthesis related infections within 1 year after TKA | 1 year
  Causes if infection are subdivided into the following:
  1. Deep prosthesis related infection
  2. Superficial infection (defined as surgery verified infection above level of the fascia)
  3. Clinical / paraclinical suspicion of infection only treated with intravenous antibiotics (no surgical procedure)
  4. Possible infection, but no clinical/paraclinical suspicion of infection, why the patient is discharged without intravenous antibiotic treatment/surgery.
  5. Surgical wound revision (no clinical/paraclinical suspicion of infection)
  6. Surgical knee manipulation due to limited range of movement (no clinical/paraclinical suspicion of infection).
  7. Surgery due to aseptic non-traumatic loosening of the knee.
  8. Surgery due to traumatic loosening of the knee

SECONDARY OUTCOMES:
Frequency and cause of hospital stay >4 days | primary admission
  Patients admitted for >4 days will have their discharge files reviewed with regards to causes of this prolonged" stay. This in accordance with the method used in the Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement registry trials (Clinicaltrials.gov identifier:NCT01515670)
Frequency and causes of 90 days readmissions | 90 days after surgery
  These will be found through review of medical files and defined as readmission possibly related to surgery and with overnight stay in hospital. These will be classified according to the method used in the ongoing trials in the Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement registry (Clin.trials ID:NCT01515670)
Frequencies and causes of readmissions to orthopedic departments 12 months after TKA. | 1 year
  These will be found through review of medical files and classified appropriately into broad categories depending on data. Detailed information on each case will be recorded
mortality | 90 days and 1 year
  Incidence of 90 days and 1 year mortality will be reported

OTHER OUTCOMES:
Prosthesis related infections 24 months after TKA | 2 years
  A separate outcome regarding incidence of prosthesis related infections, as defined in the primary outcome, is planned. This will not be part of the initial study, but is planned to be an independent follow-up study

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer C Jørgensen, MD, Principal Investigator — Section for Surgical Pathophysiology Copenhagen University, Rigshospitalet; Troels H Lunn, MD, PhD, Principal Investigator — Section for Surgical Pathophysiology, Copenhagen University, Rigshospitalet; Henrik Kehlet, MD Prof PhD, Study Chair — Secton for Surgical Pathophysiology, Copenhagen University , Rigshospitalet
Locations (7):
- Denmark (7):
  - Aarhus University Hospital, Aarhus, Judland
  - Farsoe Hospital, Farsø, Judland
  - Sydvestjydsk Sygehus, Grindsted, Judland
  - Holstebro Hospital, Holstebro, Judland
  - Vejle Hospital, Vejle, Judland
  - Viborg Hospital, Viborg, Judland
  - Gentofte University Hospital, Gentofte Municipality